CLINICAL TRIAL: NCT01829685
Title: A 3-year, Open-lable, Multi-center Extension Trial of Entecavir Therapy for Patients Previously Treated in Dragon Study
Brief Title: Efficacy Optimizing Extension Study of Chronic Hepatitis B Patients With Inadequate Response to NUC Therapy
Acronym: Dragon-Ex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China Eleventh Five-year (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-06
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis B; Inadequate Response; Nucleos(t)Ide Analogues Treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): oral entecavir 1mg daily and adefovir 10mg daily for 144 weeks
  Interventions: Drug: Entecavir, Adefovir
- Group II (Active Comparator): oral entecavir 0.5mg daily and adefovir 10mg daily for 144 weeks
  Interventions: Drug: Entecavir, Adefovir

INTERVENTIONS:
Drug: Entecavir, Adefovir

SUMMARY:
The purpose of this study is to compare the long-term efficacy and safety of entecavir 1.0 mg/d + adefovir 10 mg/d with entecavir 0.5 mg/d + adefovir 10 mg/d for chronic hepatitis B patients with inadequate response to NUC therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the 104-week Dragon study.
* Subjects who are willing to participate the extension study.

Exclusion Criteria:

* Subjects who could not compliance with the protocol judged by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Percentages of patients achieving HBV DNA< 300copies/mL at week 144 in each group | Week 144

SECONDARY OUTCOMES:
Percentages of patients achieving HBV DNA <300copies/mL at week 48/96 in each group. | Week 48 & 96
The log10 reduction in HBV DNA from baseline of DRAGON study at week 48/96/144. | Week 48 & 96 &144
Percentage of patients with HBeAg loss or HBeAg seroconversion at week 48/96/144. | Week 48 & 96 & 144
Percentage of patients with ALT normalization at week 48/96/144 | Week 48 & 96 & 144

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (16):
- China (16):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached To The Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People's Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Department of Infectious Disease, Nanfang Hospital, Guangzhou, Guangdong
  - GuangDong Provincial People's hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shengyang, Liaoning
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Li Y, Pan CQ, Ji S, Yan G, Cheng J, Liu S, Xing H. Serum IL-21 levels predict HBeAg decline during rescue therapy in patients with partial response to nucleos(t)ide analogues. Exp Ther Med. 2021 Mar;21(3):216. doi: 10.3892/etm.2021.9648. Epub 2021 Jan 15. PMID 33500704